CLINICAL TRIAL: NCT06932536
Title: A Randomized, Double-blind, Placebo-controlled Phase I Bridging Study to Evaluate the Pharmacokinetics, Safety and Tolerability of SR750 (Formulation F1) in Chinese Healthy Subjects
Brief Title: The Pharmacokinetics (PK), Safety, Tolerability of SR750 (Formulation F1) in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai SIMR Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: SR750-103
Record Dates: First submitted 2025-04-10; First posted 2025-04-17 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SR750 tablet (Experimental): Ascending single (30-100 mg) and multiple (30-60 mg twice daily [b.i.d.]) doses of SR750 orally
  Interventions: Drug: SR750 tablet
- Placebo (Placebo Comparator): Ascending single and multiple doses of placebo orally
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SR750 tablet — Ascending single (30-100 mg) and multiple (30-60 mg twice daily [b.i.d.]) doses of SR750 orally
  Arms: SR750 tablet
Drug: Placebo — Ascending single and multiple doses of placebo orally
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled phase I bridging study to evaluate the PK, safety and tolerability of SR750 (formulation F1) in Chinese healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males and females who are 18 to 45 years of age.
2. Based on medical history, physical examination, laboratory examination, chest X-ray, abdominal B-ultrasound, vital signs and ECG, the investigator considered that the results were normal or abnormal but no clinical significance.
3. Bodyweight of male > 50 kg, Bodyweight of female > 45 kg and body mass index (BMI) between 18 and28 kg/m2
4. Male subjects must agree to use contraception methods.
5. Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.

Exclusion Criteria:

1. Known history of renal dysfunction or creatinine clearance < 90 mL/min (calculated using the Cockcroft-Gault formula) at Screening.
2. Current or chronic history of liver disease or known hepatic or biliary abnormalities.
3. History of regular alcohol consumption within 6 months of screening defined as: an average weekly intake of >21 units for males or >14 units for females. One unit is equivalent to 8 g of alcohol: a half-pint (~285 mL) of beer, 1 glass (125 mL) of wine or 1 measure (25 mL) of spirits.
4. History of significant drug abuse within one year of screening or use of soft drugs (such as marijuana) within 3 months prior to screening or hard drugs (such as cocaine, methamphetamine, crack) within 1 year prior to screening.
5. History of sensitivity to any of the investigational medicinal products (IMPs), or components thereof or a history of drug or other allergy that, in the opinion of the Investigator or Medical Monitor, contraindicates participation.
6. History of asthma (excluding resolved childhood asthma), severe allergic responses.
7. History of hypercoagulable state or history of thrombosis.
8. A positive Hepatitis B surface antigen, positive Hepatitis C antibody and positive test for human immunodeficiency virus (HIV) antibody.
9. Within 6 months of screening, Smoking more than 4 cigarettes per day (including e-cigarettes).
10. A positive drug/alcohol result at Screening or Day -1.
11. Donation or lost in excess of 500 mL of blood within 56 days of Day 1 or donation of plasma within 14 days of Day 1.
12. The subject has participated in a clinical trial within 3 months of receiving IMP.

    Use of medication other than topical products without significant systemic absorption.
13. Unable to refrain from consumption of Seville oranges, grapefruit or grapefruit juice within 24h prior to the first dose of IMP until the Safety Follow-up visit.
14. Female subjects with positive pregnancy test results.
15. The investigator will determine any conditions in which subjects are not suitable for the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2025-04-28 (Actual); Primary Completion 2025-07-07 (Actual); Study Completion 2025-07-07 (Actual)

PRIMARY OUTCOMES:
Cmax | Up to 48 hours post-dose
  Peak plasma concentration
Tmax | Up to 48 hours post-dose
  Time of peak plasma concentration
AUC | Up to 48 hours post-dose
  Area under the plasma concentration-time curve
CL/F | Up to 48 hours post-dose
  Apparent oral clearance
t1/2 | Up to 48 hours post-dose
  Terminal half-life
Rac | Up to 48 hours post-dose
  Accumulation ratio

SECONDARY OUTCOMES:
AE: Adverse Event | Up to Day 7(+ 7 days) for the safety follow up post-dose
  The frequency and severity of althy volunteers administrated with single and repeated oral doses of SR750 AEs

CONTACTS AND LOCATIONS:
Overall Officials: Qian Chen, Principal Investigator — Shanghai Clinical Research Center Phase I Clinical Research Unit (SCRC-PCRU)
Locations (1):
- Shanghai Clinical Research Center Phase I Clinical Research Unit (SCRC-PCRU), Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No